CLINICAL TRIAL: NCT03713203
Title: An Interventional, Phase II, Non Randomized, Mono-centric Study on the Clinical Efficacy and Safety of the Medical Device PAGETEX® as a Photodynamic Therapy Device in the Treatment of Extra-Mammary Paget's Disease of the Vulva (EMPV)
Brief Title: PAGETEX® Photodynamic Therapy Device for the Treatment of Extra Mammary Paget's Disease of the Vulva (EMPV).
Acronym: PAGETEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Galderma R&D (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017_71; 2018-A01873-52 (Other: ID-RCB number, ANSM); 2018-002604-13 (EudraCT Number)
Record Dates: First submitted 2018-10-15; First posted 2018-10-19 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Paget Disease of the Vulva; Paget Disease, Extramammary
Keywords: Photodynamic Therapy (PDT); Medical Device; Paget Disease; Metvixia®
MeSH Terms: conditions — Paget Disease, Extramammary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pagetex PDT (Experimental): PAGETEX medical device for photodynamic therapy (PDT). Composed of the association: "Laser source + optical fiber + diffuser support incorporating luminous textiles + drug photosensitizer (Metvixia®)"
  Interventions: Device: pagetex PDT

INTERVENTIONS:
Device: pagetex PDT — 2 to 4 sessions of PDT treatment during 2.5 hours after application of Metvixia and incubation under occlusive coat.

SUMMARY:
Vulvar Paget's disease is a rare skin tumour which affect Caucasian post-menopausal women. The disease is revealed by erythematous, eczematous, pruritus and vulvar burns. The diagnosis is often late (from a few months to several years) because the symptoms are neglected by patients or misinterpreted by doctors. The reference treatment is based on surgical excision but unfortunately local recurrences are very frequent (17 to 38% of cases).

Photodynamic therapy (PDT) is already used in some dermatological pathologies and could therefore be an alternative treatment.

The objective of this study is to assess the efficacy and evaluate the safety of the new PDT device "PAGETEX" for the treatment of vulvar Paget's disease.

ELIGIBILITY:
Inclusion Criteria:

* Non-invasive, primary or recurrent vulvar Paget's disease after surgical resection
* Ability to give informed consent.
* Ability to adhere to the study protocol
* Patients must have biopsy (< 1year) proven recurrent extra mammary Paget's disease
* Effective contraception for Women of childbearing potential

Exclusion Criteria:

* Invasive vulvar Paget's Disease
* Underlying adenocarcinoma
* Subject to photosensitive disorders / reactions
* Treatment with Imiquimod / Aldara 5% cream in the last 3 months
* Photodynamic therapy used to treat MPV lesions in the last 3 months
* Use of photosensitive agents in the last 3 months
* Treatment with an experimental drug in the 30 days prior to the start of the study,
* Allergic or hypersensitivity to methyl aminolevulinate or any of the other ingredients of this medication (propyl p-hydroxybenzoate, cetostearyl alcohol, methyl p-hydroxybenzoate)
* Allergic or hypersensitivity to peanut or soya due to the presence of peanut oil in Metvixia®
* Patient with Porphyria
* Patient already treated with topical corticosteroids on the injured area in the last 3 months
* Patients with immunity disorders (HIV, transplantation)
* Clinical follow-up impossible for psychological, family, social or geographical reasons,
* Legal incapacity
* Pregnant or lactating woman
* Refuse to participate in or sign the consent of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients diagnosed with Paget's Disease Extra-Mammary Vulvae confirmed by biopsy of less than one year.
Enrollment: 24 (Estimated)
Dates: Start 2019-08-27 (Actual); Primary Completion 2026-08-27 (Estimated); Study Completion 2026-08-27 (Estimated)

PRIMARY OUTCOMES:
disease control rate in 30% of patients included | At 3 months
  Clinical response will be assessed by vulvar examination by the investigator and independent medical committee. Measurement is defined as complete remission, partial remission (decrease by >50% of total lesion size), stability ( decrease by <50% of total lesion size )or progression of the disease

SECONDARY OUTCOMES:
disease control rate in 30% of patients included | at 6 months
  Clinical response will be assessed by vulvar examination by the investigator and independent medical committee. Measurement is defined as complete remission, partial remission (decrease by ≥50% of total lesion size), stability ( decrease by <50% of total lesion size )or progression of the disease
Subject discomfort measured during each treatment using a Visual Analogic Scale Evaluation of pain | At session 1 and session 2, spaced 15 day; and at session 3 and session 4 spaced 15 days (sessions 3 ; 4 in case of persistent lesions)
  Visual Analogic Scale Evaluation of pain (0 = no pain to 10= unbearable)
Clinical Evolution measured using an erythema 4 points scale and Chroma meter CR400 measures | at 3 months, at 6 months
  erythema 4 points scale (0 = no erythema, 3=severe erythema) and Chroma meter CR400 (Konica Minolta) measures
Presence/absence of Paget cells in vulvar biopsy. | at 3 months, at 6 months
Change in score Dermatology Life Quality Index (DLQI) | at 3 months, at 6 months
  DLQI is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person The scoring of each question is as follows:Very much/A lot/A little/Not at all/Not relevan
Change in SF 36 | at 3 months, at 6 months
Change in Hospital Anxiety and Depression Scale. (HADS) | at 3 months, at 6 months
  Each item on the questionnaire is scored from 0-3
Change in The Female Sexual Function Index (FSFI) | at 3 months, at 6 months
  The FSFI is a brief questionnaire measure of sexual functioning in women. 19 questions scoring as follow : 0 = Did not attempt intercourse ;1 = Almost always or always 2 = Most times (more than half the time);3 = Sometimes (about half the time);4 = A few times (less than half the time); 5 = Almost never or never
Presence or absence of fluorescence on the Dermoscope Fotofinder® photographs | at 6 months
number of Adverse Events | during the study period, an average 6 months
  Incidence and severity of adverse device effects during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Mortier, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Claude Huriez, CHU, Lille, France

REFERENCES:
- [Derived] Lecomte F, Thecua E, Ziane L, Deleporte P, Duhamel A, Maire C, Staumont-Salle D, Mordon S, Mortier L. Photodynamic Therapy Using a New Painless Light-Emitting Fabrics Device in the Treatment of Extramammary Paget Disease of the Vulva (the PAGETEX Study): Protocol for an Interventional Efficacy and Safety Trial. JMIR Res Protoc. 2019 Dec 3;8(12):e15026. doi: 10.2196/15026. PMID 31793891